CLINICAL TRIAL: NCT00473551
Title: Anti-Third Party T Lymphocytes With Nonmyeloablative Stem Cell Transplantation for Treatment of Indolent Lymphoid Malignancies
Brief Title: Anti-Third Party T Lymphocytes With Nonmyeloablative Stem Cell Transplantation for Indolent Lymphoid Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0682
Record Dates: First submitted 2007-05-11; First posted 2007-05-15 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-12

CONDITIONS: Leukemia; Lymphoma; Myeloma
Keywords: Chronic Lymphocytic Leukemia; Lymphoma; Myeloma; Leukemia; Anti-Third Party Cytolytic Lymphocytes; Indolent Lymphoid Malignancies; Fludarabine; Fludara; Rituximab; Rituxan; Cyclophosphamide; Cytoxan®; Neosar®; Stem Cell Transplantation; T-lymphocytes; Miltenyi CliniMACS System; Graft vs. Host Disease; GVHD; Allogenic Transplant; Sirolimus; Rapamycin
MeSH Terms: conditions — Leukemia; Lymphoma; Neoplasms, Plasma Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Graft vs Host Disease | interventions — Rituximab; Cyclophosphamide; fludarabine; fludarabine phosphate; Mesna; Radiotherapy; Stem Cell Transplantation; Sirolimus; Lymphocyte Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anti-Third Party T Lymphocytes + Nonmyeloablative SCT (Experimental): Anti-Third Party CTL (Cytolytic T-lymphocytes) with Nonmyeloablative SCT (Stem Cell Transplantation)
  Rituximab 375 mg/m^2 intravenously over several hours on Day -13, followed by 1000 mg/m^2 intravenously on Days -6, 1, and 8; + Cyclophosphamide 50 mg/kg intravenously over two hours on Day -6, immediately following Fludarabine; + Fludarabine 40 mg/m^2 intravenously over 30 minutes once per day for 4 days, starting Day -6; + Radiation 2Gy Total body radiation day before transplantation + Stem Cell Transplantation + Intravenous infusion of Anti-third Party CTLs.
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Mesna; Radiation: Radiation Treatment; Procedure: Stem Cell Transplantation (SCT); Drug: Sirolimus; Procedure: Anti-third Party Cytolytic T-lymphocytes (CTL)

INTERVENTIONS:
Drug: Rituximab — 375 mg/m^2 intravenously over several hours on Day -13, followed by 1000 mg/m^2 intravenously on Days -6, 1, and 8.
  Other Names: Rituxan
Drug: Cyclophosphamide — 50 mg/kg intravenously over two hours on Day -6, immediately following Fludarabine.
  Other Names: Cytoxan®; Neosar®
Drug: Fludarabine — 40 mg/m^2 intravenously over 30 minutes once per day for 4 days, starting Day -6.
  Other Names: Fludarabine Phosphate; Fludara
Drug: Mesna — 10 mg/kg continuous intravenous infusion for 4 hours for total of 6 doses (24 hours) following Cyclophosphamide.
Radiation: Radiation Treatment — 2Gy Total body radiation day before transplantation
  Other Names: XRT; RT; Radiotherapy
Procedure: Stem Cell Transplantation (SCT) — Allo CD34+ Selected SCT/Infusion of stem cells.
  Other Names: Nonmyeloablative Stem Cell Transplantation
Drug: Sirolimus — 6 mg by mouth on day -2 followed by 2 mg daily from day -1 through day +7.
  Other Names: Rapamycin
Procedure: Anti-third Party Cytolytic T-lymphocytes (CTL) — Intravenous infusion of anti-third party CTL.
  Other Names: Third Party T-Cells; Lymphocytes

SUMMARY:
Primary Objective:

1. To determine the maximally tolerated dose of anti-third party cytolytic T-lymphocytes, defined as the dose which achieve engraftment without severe GVHD (graft-vs-host disease) at 90 days after allogeneic transplantation of CD34+ hematopoietic progenitor cells.

Secondary Objective:

1. Toxicity, response rate, time to progression and overall survival.

DETAILED DESCRIPTION:
GVHD can be a major problem after stem cell transplantation from a healthy donor. It is caused by T-lymphocytes (a type of immune cell) from the donor that can react badly against the person receiving the transplant (the recipient). Researchers want to see if stimulating the donor T-lymphocytes against another person (a third party) and growing them for 28 days will decrease the chance of developing GVHD.

If you are found to be eligible to take part in this study, you will receive the below treatment, including chemotherapy and radiation, before your stem cell transplantation. These include rituximab, cyclophosphamide, fludarabine, and mesna. Rituximab is designed to attach to lymphoma cells, causing them to die. Cyclophosphamide is designed to destroy cancer cells by interfering with their multiplication and slowing or stopping their growth and spread throughout the body. Fludarabine is designed to interfere with DNA repair enzymes so that the leukemic cell cannot repair damaged DNA. This increases the likelihood of the cell dying. Mesna is a drug that lowers the risk of bladder side effects by the cyclophosphamide. Total body radiation is given to to reduce the risk of transplant rejection.

Participants with CLL or lymphoma will receive Rituxan (rituximab) by vein, given over several hours for each dose. The first rituximab dose is 13 days before the transplant. This will be followed by 3 more doses of rituximab, given 6 days before the transplant, and 1 and 8 days after the transplant. All participants will receive fludarabine by vein over 30 minutes once per day for 4 days, starting 6 days before the transplant. All participants will also receive cyclophosphamide by vein over 2 hours. The cyclophosphamide will be given immediately after the first dose of fludarabine. All participants will also receive a continuous infusion of mesna by vein for 24 hours after receiving the cyclophosphamide. One day before transplantation, you will have total body radiation.

After receiving total body radiation, you will receive your stem cell transplantation. On the day of the transplant, you will receive the anti-third party T Lymphocytes (CTLs) by vein. This will be followed by vein infusion of stem cells from the donor. A sample of the anti-third party T-cells cells will also be tested for immune function.

All participants will receive sirolimus by mouth for 10 days, starting 2 days before transplantation. Sirolimus is an immunosuppressive drug which is given to reduce the risk of transplant rejection. You will remain in the hospital for about 4 weeks after the transplant. You will then continue as an outpatient in the Houston area for 100 days after your transplantation, or until your doctor feels it is okay for you to leave the Houston area.

If your disease gets worse after your transplantation, you may receive additional immune cells from the donor (DLI-donor lymphocyte infusion).You may be taken off this study if the transplant does not grow or is rejected, if not enough of the CTLs can be produced, if your disease continues to get worse after receiving additional donors cells, or if you experience any intolerable side effects.

You will have frequent blood tests as medically necessary to evaluate your medical condition. About 3 tablespoons of blood will be collected for immune function testing at 1, 2, 3, 6 and 12 months after the transplant. You will have a bone marrow biopsy, x-rays, and CT scans for evaluation of the cancer at 1, 3, 6, 9, and 12 months after the transplant. The study is over after 1 year. You will be followed-up after that time for routine care, as the doctors feels it is necessary.

This is an investigational study. All of the drugs used in this study, have been approved by the FDA in the treatment of cancer and transplantation. The Miltenyi CliniMACS System which is used to purify stem cells and the anti-third party CTLs has not been approved by the FDA, and its use in this study is experimental. Up to 24 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* Confirmed diagnosis of follicular lymphoma, mantle cell lymphoma, chronic lymphocyte leukemia/small lymphocytic lymphoma or multiple myeloma. Patients must have had persistent or progressive disease despite initial chemotherapy. Patients must have achieved a partial or complete response to their most recent chemotherapy.
* Patients must have an human leukocyte antigen (HLA) matched (HLA-A, B, C DR or DQ) related donor who is seropositive against Epstein Barr virus and capable of donating peripheral blood mononuclear cells and peripheral blood progenitor cells.
* Patient must be HLA completely mismatched for HLA class I loci (A, B and C) with the 3rd party stimulator cells. HLA-A (330301, 310102) HLA-B (5801,150101[62]) HLA-C (0302, 030301)
* Zubrod Performance Scale (PS) of 0 or 1
* Creatinine < 1.8 mg/dl
* Ejection fraction >/=40%
* Corrected Carbon Monoxide Diffusing Capacity (DLCO) >/=45% predicted
* Serum bilirubin </=1.5 mg/dl if not due to Gilbert's syndrome

Exclusion Criteria:

* Uncontrolled infection
* HIV, hepatitis B surface antigen or hepatitis C seropositive
* serum glutamic-pyruvic transaminase (SGPT) > 200 IU/ml
* Pregnant or lactating women i.e., positive Beta human chorionic gonadotrophin (hCG) test in a woman with child bearing potential. Child bearing potential is defined as not post-menopausal for 12 months or no previous surgical sterilization.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-05; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants achieving engraftment without severe Graft-versus-host disease (GVHD) | Baseline to 90 days
  Number of participants who achieve engraftment without severe GVHD at 90 days after allogeneic transplantation of CD34+ hematopoietic progenitor cells. Engraftment recorded as first day of three (3) consecutive days that the Absolute neutrophil count (ANC) exceeds 0.5 * 109/L. Graft failure is defined as failure to reach an ANC > 0.5 * 109/L within 28 days after transplantation with detectable donor cells on chimerism analysis.
Maximally tolerated dose of anti-third party cytolytic T-lymphocytes | Baseline to 90 days
  Maximally tolerated dose of anti-third party cytolytic T-lymphocytes, defined as the dose which achieve engraftment without severe GVHD at 90 days after allogeneic transplantation of CD34+ hematopoietic progenitor cells. Engraftment recorded as first day of three (3) consecutive days that the Absolute neutrophil count (ANC) exceeds 0.5 * 109/L. For dose-finding, "toxicity" is defined as either death or acute GVHD (aGVHD) within 90 days and "response" is defined as the event the patient is alive and engrafted at day 30.

CONTACTS AND LOCATIONS:
Overall Officials: Richard E. Champlin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center website — http://www.mdanderson.org